CLINICAL TRIAL: NCT05780450
Title: Effectiveness of Transcranial Direct Current (tDCS) Treatment in Patients With Persistent Covid Who Present Headaches and Chronic Body Pain.
Brief Title: Effectiveness of Transcranial Direct Current in Patients With Persistent COVID-19 With Headaches and Chronic Pain.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCV/2021-2022/140
Record Dates: First submitted 2023-03-13; First posted 2023-03-22 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; Long COVID; Long Covid19; SARS CoV 2 Infection; Persistent COVID-19; Migraine Disorders; Headaches Chronic; Cluster Headache; Arthralgia; Myalgia; Chronic Pain; Post-COVID-19 Syndrome; Post COVID-19 Condition
Keywords: Transcranial Direct Current Stimulation; tDCS; Covid Persistente
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome; Migraine Disorders; Headache Disorders; Cluster Headache; Arthralgia; Myalgia; Chronic Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental)
  Interventions: Device: Transcranial Direct Current Therapy (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Therapy (tDCS) — Transcranial direct therapy (tDCS) is a non-invasive neuromodulation therapy of the cerebral cortex, which consists of the application of electrical microcurrents, of approximately 2mA, through surface electrodes placed on the scalp. Transcranial therapy (tDCS) produces immediate effects on the ability of neurons to change their electrical potential.
  Each session lasts between 20 and 30 minutes, and approximately 10 consecutive sessions should be performed. It will be applied through two surface electrodes of 25 to 35 cm2 at 2 mA.
  The equipment has a European health certificate (CE), so it is an approved equipment that complies with all the safety measures for the application of the treatment.

SUMMARY:
This study aims to verify the efficacy / effectiveness of treatment with transcranial direct therapy (TDCS) in patients with Persistent Covid who present headaches, migraines and chronic pain, such as arthralgias and myalgias.

Transcranial Direct Therapy is used in the field of Physiotherapy and Rehabilitation, with results that prove to be effective for the treatment of patients suffering from symptoms such as migraines, headaches, chronic pain, fibromyalgia or chronic neuropathic pain.

As can be seen, in the case of patients with Persistent Covid we find several of these symptoms, so it is suggested that, if Transcranial Direct Current Therapy (TDCs) is giving such good results, relieving these symptoms, why can not give such good results and help so much in patients with Persistent Covid, If many of the symptoms are the same, even if the origin or cause is different.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Persistent Covid
* Men and women
* All ages from 16 years old
* Patients who passed the Covid in its acute phase in an asymptomatic, mild and severe way.

Exclusion Criteria:

* Patients without confirmation with positive PCR in the acute phase of Covid-19
* Patients with Persistent Covid who do not have at least one of these symptoms: migraines, headaches, chronic pain, neuropathic pain, arthralgia, myalgias
* Patients with pacemaker / defibrillator
* Patients with brain implants
* Patients with cranial fractures
* Pregnant

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
CHANGE FROM PRE-TREATMENT DEGREE CHRONIC BODY PAIN AT INMEDIATE POST-TREATMENT, 1 MONTH AND 3 MONTHS | PRE-TREATMENT / IMMEDIATE POST-TREATMENT / POST-TREATMENT 1 MONTH / 3 MONTHS
  MEASURED WITH 2 SPECIFIC PAIN SCALES (EVA-Visual Analog SCALE AND MCGILL PAIN QUESTIONNAIRE). EVA SCALE (0 no pain-10 maximun pain). MCGILL QUESTIONNAIRE (0 no pain-66 maximun pain)
CHANGE FROM PRE-TREATMENT INTENSE MIGRAINES OR HEADACHES AT INMEDIATE POST-TREATMENT, 1 MONTH AND 3 MONTHS | PRE-TREATMENT / IMMEDIATE POST-TREATMENT / POST-TREATMENT 1 MONTH / 3 MONTHS
  MEASURED WITH 2 SPECIFIC SCALES (MIDAS-Migraine dissability Assessment SCALE AND HIT-6 QUESTIONNAIRE-headache impact test). MIDAS SCALE (0 nil disability - >21 severe disability). HIT-6 QUESTIONNAIRE (0 no impact - >60 very severe impact).

SECONDARY OUTCOMES:
CHANGE FROM PRE-TREATMENT QUALITY OF LIFE (SF-12 QUESTIONNAIRE) AT INMEDIATE POST-TREATMENT, 1 MONTH AND 3 MONTHS | PRE-TREATMENT / IMMEDIATE POST-TREATMENT / POST-TREATMENT 1 MONTH / 3 MONTHS
  MEASURED WITH 1 SPECIFIC SCALE (SF-12 QUESTIONNAIRE). (0 worst quality of life - 100 best quality of life)
CHANGE FROM PRE-TREATMENT MOOD AT INMEDIATE POST-TREATMENT, 1 MONTH AND 3 MONTHS | PRE-TREATMENT / IMMEDIATE POST-TREATMENT / POST-TREATMENT 1 MONTH / 3 MONTHS
  MEASURED WITH 1 SPECIFIC SCALE (EVEA-mood rating SCALE). (0 nothing - 10 a lot)

CONTACTS AND LOCATIONS:
Overall Officials: LAURA GARCÍA MARTÍNEZ, Principal Investigator — Escuela de Doctorado. Universidad Católica de Valencia San Vicente Mártir. (Doctoral School. Catholic University of Valencia San Vicente Mártir)
Locations (2):
- Spain (2):
  - Clínica Paiporta, Paiporta, Valencia
  - Escuela de Doctorado. Universidad Católica de Valencia San Vicente Mártir. (Doctoral School. Catholic University of Valencia San Vicente Mártir), Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conde-Anton A, Hernando-Garijo I, Jimenez-Del-Barrio S, Mingo-Gomez MT, Medrano-de-la-Fuente R, Ceballos-Laita L. Effects of transcranial direct current stimulation and transcranial magnetic stimulation in patients with fibromyalgia. A systematic review. Neurologia (Engl Ed). 2020 Oct 15:S0213-4853(20)30278-4. doi: 10.1016/j.nrl.2020.07.024. Online ahead of print. English, Spanish. PMID 33071017
- [Background] Pacheco-Barrios K, Cardenas-Rojas A, Thibaut A, Costa B, Ferreira I, Caumo W, Fregni F. Methods and strategies of tDCS for the treatment of pain: current status and future directions. Expert Rev Med Devices. 2020 Sep;17(9):879-898. doi: 10.1080/17434440.2020.1816168. Epub 2020 Sep 15. PMID 32845195